CLINICAL TRIAL: NCT04560504
Title: Oculomotor Deficits in Parkinson's Disease: Enhancing Eye Movement Performance and Dynamic Visual Acuity With Oculomotor Training Using a Pilot Randomized Clinical Trial Design
Brief Title: Effectiveness of Oculomotor Training in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: University of California, Berkeley (Other); Deakin University (Other); Chinese University of Hong Kong (Other); Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Allen MY Cheong, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 15102717
Record Dates: First submitted 2020-09-07; First posted 2020-09-23 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Parkinson Disease; Oculomotor; Disorder
Keywords: Parkinson Disease; Oculomotor deficit; Oculomotor training; Dynamic vision
MeSH Terms: conditions — Parkinson Disease | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Receive 10 sessions of 45-minute (3 sessions per week) in-office leisure activities e.g. simple non-action computer games or board games (e.g. card and chess games) and 10-20 minutes of video watching at home
  Interventions: Other: Control Group
- Intervention Group (Active Comparator): Receive 10 sessions of 45-minute office training (3 sessions per week) and 10-20 minute home training (3 sessions per week) of eye movement training
  Interventions: Other: Oculomotor Training Group

INTERVENTIONS:
Other: Control Group — Leisure activities
  Arms: Control Group
Other: Oculomotor Training Group — Eye movement training
  Arms: Intervention Group

SUMMARY:
Parkinson's disease (PD) is a common neurodegenerative disorder which is characterized by both motor and non-motor symptoms and usually affects people aged 50 years or above. Many studies showed eye movement deficits and visual changes in patients with PD.

Previous studies have also indicated that clinical eye movement training could enhance the functional performance of patients with various eye movement problems resulting from ocular and neurodegenerative diseases.

In this study, we will investigate the effectiveness of eye movement training on dynamic vision and functional performance in PD patients with oculomotor deficits.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's Disease diagnosed by a neurologist or geriatrician with the range of Stage

  1 to 4 (Hoehn and Yahr Classification)
* Able to speak and comprehend Cantonese dialect
* Able to travel independently

Exclusion Criteria:

* Any congenital eye problem (e.g. congenital strabismus or amblyopia in either eye) or any manifest eye diseases (e.g. macular degeneration, glaucoma, etc)
* Severe medical problems (e.g. stroke)
* Cognitive impairment (e.g. dementia)
* Presence of any psychiatric or neurological diseases (apart from Parkinson's disease) or receiving of any psychoactive pharmacological treatment
* Receiving any medication that is known to affect eye movement and cognitive function
* Previous formal vision rehabilitation or oculomotor intervention

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Smooth Vergence eye movements | Change from baseline at week 4 and change from baseline at week 12
  Smooth vergence eye movement is measured using a head-mounted eye tracking while fixating at an approaching target moving at different speeds

SECONDARY OUTCOMES:
Oculomotor characteristics | Change from baseline at week 4 and change from baseline at week 12
  With the use of eye tracking device, eye movement behavior of participants can be measured and analysed while performing the following tasks.
  1. Fixation task - Fixate at stationary target presented on a monitor
  2. Saccade task - Follow and fixate at a random jumping target presented on a monitor
  3. Pursuit task - Follow accurately and steadily on a smooth moving target presented on a monitor
  4. Jump Vergence task - Follow and fixate a jumping target presented in the anterior-posterior plane (jumping from 'far to near' or 'near to far')
Sentence reading performance | Change from baseline at week 4 and change from baseline at week 12
  To evaluate the effectiveness of the interventions on sentence reading using MNREAD charts in Chinese. These charts developed in our laboratory are used to measure the effectiveness of sentence reading in terms of reading speed and critical print size.
Passage reading performance | Change from baseline at week 4 and change from baseline at week 12
  To evaluate the effectiveness of the interventions on passage reading using International Reading speed Test (IReST). IReST is used to evaluate the effectiveness of passage reading performance by measuring the reading speed.

CONTACTS AND LOCATIONS:
Overall Officials: Allen Ming Yan Cheong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Allen MY Cheong, Hong Kong, Hong Kong